CLINICAL TRIAL: NCT03327116
Title: Evaluation of the Effect of Methotrexate on Cytokines and Chemokines Involved in the Inflammatory Response in Adult Patients With Atopic Dermatitis
Brief Title: Effect of Methotrexate on Inflammatory Response in Adult Atopic Dermatitis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: FUNADERSP (Foundation for Research Support of the State of São Paulo) (Unknown)
Responsible Party: Principal Investigator, Valéria Aoki, Associate Professor and Director of International Relations, University of Sao Paulo General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13.368
Record Dates: First submitted 2017-07-30; First posted 2017-10-31 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; pruritus; methotrexate; inflamation; IL-31
MeSH Terms: conditions — Dermatitis, Atopic; Pruritus | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Methotrexate (Experimental)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Methotrexate — oral, 15 mg per week, 24 weeks

SUMMARY:
Atopic dermatitis (AD) is a chronic inflammatory skin disease associated with pruritus. Methotrexate can be used to treat refractory disease to conventional therapy.

It will be conducted a single arm trial with twelve adult patients with moderate to severe AD on methotrexate for 24 weeks.

Investigators intend to evaluate the effect methotrexate on cytokines and chemokines involved in the inflammatory response, on IgE levels, on pruritus, and on EASI and SCORAD severity scores.

DETAILED DESCRIPTION:
Introduction: Atopic dermatitis (AD) is a chronic inflammatory skin disease associated with pruritus. Methotrexate (MTX) can be used to treat refractory disease to conventional therapy, but there are few studies showing its effect on the profile of cytokines involved in the inflammatory response.

Objectives: To assess the effect of MTX on the cytokines involved in the inflammatory response of adult AD patients treated with methotrexate for 24 weeks. As specific objectives, investigators intend to assess the evolution of serum IgE levels, the EASI (Eczema Area and Severity Index) and SCORAD (Scoring Atopic Dermatitis) severity scores and pruritus in them.

Methods: It will be conducted an open, prospective study with twelve adult patients with moderate to severe AD on MTX for 24 weeks. Each participant is expected to attend 7 visits during 6 months of follow-up. In clinical healthy and injured skin, two assessments will be performed: 1) mRNA expression of IL-4, IL-10, IL-17A, IL-22, IL-31, oncostatin M receptor (OSMR), alpha subunit IL-31 (IL-31RA) receptor, TNF-α, IFN-γ, TSLP, TARC and MDC by Real Time-PCR at the initial week and week 24; 2) expression of IL-31, IL-31RA, OSMR, TSLP and Ki67 by immunohistochemistry at the initial week and week 24.

Skin samples from non-atopic subjects will be utilized as controls for the assays, paired by gender and age.

Additional analysis of serum levels of IgE (nephelometric method) at the initial week and week 24 of the study will be performed.

AD severity scores (EASI and SCORAD) will be tested and pruritus will be analyzed by a visual analog scale at the initial, week 12 and week 24.

ELIGIBILITY:
Inclusion Criteria:

* AD (Hanifin and Rajka criteria) moderate to severe (EASI ≥ 7.1 and SCORAD ≥ 25);
* Age ≥ 18 years;
* Women without the potential to become pregnant or using an effective method of contraception and with a negative pregnancy blood test;
* Men without a desire of pregnancy and who use condom in sexual intercourse.

Exclusion Criteria:

* Hepatic and / or renal insufficiency;
* Anemia, thrombocytopenia and / or leukopenia;
* Use of concomitant hepatotoxic drug;
* Active infection;
* Allergy to MTX;
* Excessive alcohol intake;
* Difficulty to understand how to take methotrexate;
* HIV infection or other immunosuppression condition;
* Therapy with UVA or UVB, corticoid, cyclosporine, immunobiological, azathioprine within 12 weeks prior to introduction of methotrexate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline of cytokines and chemokines expression at 24 weeks | week 24
  mRNA expression of IL-4, IL-6, IL-10, IL-31, TSLP, INF-gamma, TNF-alpha, TARC and MDC by Real Time-PCR.
  Immunohistochemistry with antibodies against IL-31, IL-31RA, OSMR, TSLP and Ki67

SECONDARY OUTCOMES:
Change from baseline of IgE level at 24 weeks | week 24
  Nephelometric method
Change from baseline of Pruritus at 12 weeks | week 12
  Visual analogue scale (VAS). The VAS was used as a 10-cm long horizontal line with a starting point as "no itch" (0 points) and ending with "worst imaginable itch".
Change from baseline of Pruritus at 24 weeks | week 24
  Visual analogue scale (VAS). The VAS was used as a 10-cm long horizontal line with a starting point as "no itch" (0 points) and ending with "worst imaginable itch".
Change from baseline of SCORAD severity score at 12 weeks | week 12
  The SCORAD (Scoring atopic dermatitis) is a severity score used for atopic dermatitis.
  To measure the extent of AD, the rule of nines is applied on a front/back drawing of the patient's inflammatory lesions. The extent can be graded from 0 to 100.
  The intensity part of the SCORAD consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness. Each item can be graded on a scale from 0 to 3.
  The subjective items include daily pruritus and sleeplessness. The SCORAD Index formula is: A/5 + 7B/2 + C. In this formula, A is defined as the extent (0-100), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The minimal score of SCORAD is 0 and the maximal score is 103 (most severe).
Change from baseline of SCORAD severity score at 24 weeks | week 24
  The SCORAD (Scoring atopic dermatitis) is a severity score used for atopic dermatitis.
  To measure the extent of AD, the rule of nines is applied on a front/back drawing of the patient's inflammatory lesions. The extent can be graded from 0 to 100.
  The intensity part of the SCORAD consists of 6 items: erythema, oedema/papulation, excoriations, lichenification, oozing/crusts and dryness. Each item can be graded on a scale from 0 to 3.
  The subjective items include daily pruritus and sleeplessness. The SCORAD Index formula is: A/5 + 7B/2 + C. In this formula, A is defined as the extent (0-100), B is defined as the intensity (0-18) and C is defined as the subjective symptoms (0-20). The minimal score of SCORAD is 0 and the maximal score is 103 (most severe).
Change from baseline of EASI severity score at 12 weeks | week 12
  Eczema Area and Severity Index (EASI) is a tool for the measurement of severity of atopic dermatitis.
  It ranges from 0 (no eczema) to 72 (most severe).
  EASI is one of the core outcome instruments recommended to be included in all clinical trials on atopic dermatitis.
Change from baseline of EASI severity score at 24 weeks | week 24
  Eczema Area and Severity Index (EASI) is a tool for the measurement of severity of atopic dermatitis.
  It ranges from 0 (no eczema) to 72 (most severe).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital das Clínicas of the University of São Paulo Medical School, Department of Dermatology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Samorano LP, Manfrere KCG, Pereira NV, Takaoka R, Valente NYS, Sotto MN, Silva LFF, Sato MN, Aoki V. Methotrexate for refractory adult atopic dermatitis leads to alterations in cutaneous IL-31 and IL-31RA expression. An Bras Dermatol. 2024 Jan-Feb;99(1):72-79. doi: 10.1016/j.abd.2023.01.002. Epub 2023 Sep 18. PMID 37730501